CLINICAL TRIAL: NCT06550232
Title: The Effect of IV PAPAVERINE 80 mg Prior to Propess on Bishop Score and Pain, Double Blinded Randomized Placebo Controlled Trial
Brief Title: IV PAPAVERINE Prior to Propess for Labor Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Head of Fetal Maternal Unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0112-24-NHR
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Induced Vaginal Delivery
Keywords: labor induction; papaverine; propess; bishop score; induction to delivery interval
MeSH Terms: interventions — Papaverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group allocation will be double blind. The randomization table will be available only to one member of the study, who will prepare the medications according to the allocated intervention. Participants will receive intravenous 0.9% normal saline with or without papaverine. The same bottles of normal saline will be use for the papaverine and placebo groups. Accordingly, the participants will be masked for the intervention. The participants, the researchers including the obstetricians who inserted the PGE2 (propess), the caregiver nurse who administrated the medication, the data collector, and the statistician will be blinded to the group allocations throughout the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- papaverine arm (Active Comparator): IV-papaverine 80 mg in 100 ml 0.9% saline, once
  Interventions: Drug: Papaverine
- Control arm (Placebo Comparator): I.V 100 ml 0.9% saline
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Papaverine — Within 30-minutes prior to catheter insertion, women in the intervention group will receive IV-papaverine 80 mg in 100 ml 0.9% saline
  Arms: papaverine arm
Other: placebo — I.V Sallne
  Arms: Control arm

SUMMARY:
The investigators aim to evaluate the effect of administering papaverine prior to PGE2 insertion on changes in Bishop-scores and on the induction-to-delivery interval.

Researchers will compare drug papaverine to a placebo

DETAILED DESCRIPTION:
More than 22% of all pregnant women undergo induction of labor. Induction of labor is usually medically indicated for maternal and fetal related conditions; however, elective induction has become more common since the ARRIVE trial. Women with an unfavourable cervix, according to Bishop-score (<6), are prone to higher induction failure rates and are candidates for cervical ripening.

The cervix is composed of connective tissue and smooth-muscle located mainly beneath the internal os. Papaverine is an antispasmodic-musculotropic drug that targets smooth-muscle, resulting in decreased muscle spasm and subsequent smooth-muscle relaxation. The half-life of the drug is in the range of 0.5-2 hours, and its action starts 10 minutes after administration. Short-term use of papaverine during the first trimester has been reported as safe. However, outcome data are lacking of the use of mucosotropic-agents prior to PGE2 (propess) insertion. We will investigate this in a trial in which the co-primary outcomes were the change in Bishop-score after PGE2 extraction and the PGE2 insertion-to-delivery interval

ELIGIBILITY:
Inclusion Criteria:

* singleton term pregnancy
* bishop score
* need for labor induction with PGE2
* vertex presentation
* viable fetus

Exclusion Criteria:

* Prelabour rupture of membrane
* Twins pregnancy
* previous cesarean section
* allergy to the study medication
* fetal anomaly contraindications for vaginal delivery
* maternal supraventricular tachicardia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 110 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Delta Bishop score | 24 hours
  The bishop score before and after propess insertion
the time from propess insertion until delivery | 72 hours
  induction to delivery time

SECONDARY OUTCOMES:
maternal satisfaction scores | 24 hours
  maternal satisfaction on 1-5 scale. higher scores mean higher satisfaction
visual analogue scale score | 24 hours
  pain assessment using a 10-point visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Yes
The authors are willing to share the data of the study upon request of the Editors.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Oliveira MV, Oberst PV, Leite GK, Aguemi A, Kenj G, Leme VD, Sass N. [Cervical Foley catheter versus vaginal misoprostol for cervical ripening and induction of labor: a randomized clinical trial]. Rev Bras Ginecol Obstet. 2010 Jul;32(7):346-51. doi: 10.1590/s0100-72032010000700007. Portuguese. PMID 21152844
- [Background] Rohwer AC, Khondowe O, Young T. Antispasmodics for labour. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD009243. doi: 10.1002/14651858.CD009243.pub2. PMID 22895986
- [Background] Singh KC, Jain P, Goel N, Saxena A. Drotaverine hydrochloride for augmentation of labor. Int J Gynaecol Obstet. 2004 Jan;84(1):17-22. doi: 10.1016/s0020-7292(03)00276-5. PMID 14698825
- [Background] Ibrahim MI, Alzeeniny HA, Ellaithy MI, Salama AH, Abdellatif MA. Drotaverine to improve progression of labor among nulliparous women. Int J Gynaecol Obstet. 2014 Feb;124(2):112-7. doi: 10.1016/j.ijgo.2013.08.013. Epub 2013 Nov 7. PMID 24299975
- [Background] Madhu C, Mahavarkar S, Bhave S. A randomised controlled study comparing Drotaverine hydrochloride and Valethamate bromide in the augmentation of labour. Arch Gynecol Obstet. 2010 Jul;282(1):11-5. doi: 10.1007/s00404-009-1188-8. Epub 2009 Jul 31. PMID 19644697
- [Background] Yilmaz B, Kart C, Kelekci S, Gokturk U, Sut N, Tarlan N, Mollamahmutoglu L. Meperidine versus valethamate bromide in shortening the duration of active labor. Int J Gynaecol Obstet. 2009 Nov;107(2):126-9. doi: 10.1016/j.ijgo.2009.06.021. Epub 2009 Aug 6. PMID 19664769